CLINICAL TRIAL: NCT05436652
Title: A Trial of Prednisolone in Combination With SPI-62 or Placebo in Subjects With Polymyalgia Rheumatica (PMR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sparrow Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: SPI-62-CL-2003
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Polymyalgia Rheumatica
Keywords: polymyalgia rheumatica; PMR; Steroids; Prednisolone; glucocorticoid; glucocorticoids
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant
Masking Description: Drug and Placebo are masked and assigned via Interactive Response Technology (IRT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SPI-62 (Experimental): Active drug / placebo by mouth each morning for up to 4 weeks + standard of care 10mg prednisolone. Each participant will receive both placebo and active drug but will be blinded to the sequence of active drug and placebo.
  Interventions: Drug: SPI-62; Drug: SPI-62 matched placebo; Drug: Prednisolone 10mg
- SPI-62 + additional prednisolone (Experimental): Active drug / placebo by mouth each morning for up to 4 weeks + standard of care 10mg prednisolone + additional prednisolone or placebo. Each participant will receive both placebo and active drug but will be blinded to the sequence of active drug and placebo.
  Interventions: Drug: SPI-62; Drug: SPI-62 matched placebo; Drug: Prednisolone 10mg; Drug: Additional prednisolone; Drug: Additional prednisolone matched placebo

INTERVENTIONS:
Drug: SPI-62 — 11β hydroxysteroid dehydrogenase type 1 (HSD-1) inhibitor
Drug: SPI-62 matched placebo — Inactive tablets identical in appearance to SPI-62 tablets
Drug: Prednisolone 10mg — Standard of care prednisolone
Drug: Additional prednisolone — Over encapsulated prednisolone
  Arms: SPI-62 + additional prednisolone
Drug: Additional prednisolone matched placebo — Inactive capsules identical in appearance to over encapsulated prednisolone
  Arms: SPI-62 + additional prednisolone

SUMMARY:
This will be a single-blind, placebo-controlled phase 2 trial to compare prednisolone effects with and without SPI-62 in participants with PMR.

DETAILED DESCRIPTION:
This will be a single-blind, placebo-controlled phase 2 trial to compare prednisolone effects with and without SPI-62 in participants with PMR. Up to 6 cohorts of 12 participants could be recruited (12 to 72 participants). Each participant who provides consent and meets all inclusion and exclusion criteria will participate in 3 periods: a screening period up to 28 days (Day -28 to Day-1), a 4-week treatment period (Day 1 to Day 28) and a follow up Period (Day 29 to Day 56). During the 4-week treatment period for the first cohort, all participants will receive prednisolone 10mg per day for 4-weeks plus SPI-62 for 2-weeks and matching placebo for 2-weeks. For cohorts 2 through 6, the dose of prednisolone co-administered with SPI-62 could be adjusted. For cohorts 5 and 6, the dose of SPI-62 could be adjusted.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of PMR according to EULAR/ACR classification criteria
* Absence of PMR relapse based on symptoms and acute phase markers
* Daily oral prednisolone 10mg dose that will have been stable for at least 1-week at the Baseline visit and is expected to remain stable during the treatment period

Exclusion Criteria:

* Any contraindication for prednisolone administration.
* A diagnosis or any clinical features of giant cell arteritis.
* Any autoimmune disease (e.g., late-onset rheumatoid arthritis) other than PMR.
* Use of medications for treatment of PMR within specified intervals prior to the Baseline Visit other than oral prednisolone.
* Use of other medications likely to interfere with trial assessments.
* History or diagnosis of endogenous hypercortisolism.
* Any current or prior medical condition, medical or surgical therapies, or clinical trial participation expected to interfere with the conduct of the trial or the evaluation of its results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Erythrocyte sedimentation rate | Baseline to Day 28
C-reactive protein | Baseline to Day 28
Plasma fibrinogen | Baseline to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: David Katz, Study Chair — Sparrow Pharmaceuticals
Locations (10):
- Germany (6):
  - Universitätsmedizin Berlin, Medizinische Klinik mit Schwerpunkt Rheumatologie und klinische Immunologie, Berlin
  - Internistische Praxisgemeinschaft Rheumatologie Nephrologie, Erlangen
  - Hamburger Rheuma Forschungszentrum II im MVZ für Rheumatologie und Autoimmunmedizin, Hamburg
  - Katholische Kliniken Rhein-Ruhr am Marien Hospital, Universitätsklinik der Ruhr-Universität, Herne
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz
  - Praxis Prof. Dr. med. Herbert Kellner, Munich
- Poland (4):
  - NovaReuma, Bialystok
  - The University of Gdańsk, Gdansk
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Dolnośląski Szpital Specjalistyczny im. T. Marciniaka, Wroclaw

IPD SHARING:
Plan to Share IPD: No